CLINICAL TRIAL: NCT00972543
Title: A Phase IV Multicentre, Randomized Double-blind, Placebo-controlled Trial to Evaluate the Safety and Efficacy of Raptiva in the Treatment of Subjects With Moderate to Severe Chronic Plaque Psoriasis Involving Palms and/or Soles, With or Without Pustules.
Brief Title: Raptiva in Palm and Sole Psoriasis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated after the European Medicines Evaluation Agency recommended to suspend the marketing authorisation of Raptiva in the European Union
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 28861
Record Dates: First submitted 2009-09-04; First posted 2009-09-07 (Estimated); Results first posted 2010-09-02 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Plaque Psoriasis
Keywords: Moderate to severe chronic plaque psoriasis; palms and/or soles; with or without pustules
MeSH Terms: interventions — efalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Raptiva (Active Comparator): Double-blind phase, Raptiva 0.7mg/kg followed by Raptiva 1mg/kg/wk for 12 weeks.There then follows an open label extension of Raptiva 0.7mg/kg followed by Raptiva 1mg/kg/wk for a further 12 weeks
  Interventions: Biological: Efalizumab (Raptiva)
- Placebo (Placebo Comparator): Double-blind phase, Placebo for 12 weeks.There then follows an open label extension of Raptiva 0.7mg/kg followed by Raptiva 1mg/kg/wk for a further 12 weeks
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Efalizumab (Raptiva) — Double-blind phase 0.7mg/kg subcutaneously (sc), followed by 1mg/kg/wk sc for 12 weeks.
  Open label extension 0.7mg/kg sc Raptiva followed by 1mg/kg/wk sc for a further 12 weeks.
  Other Names: Raptiva
  Arms: Raptiva
Biological: Placebo — Double-blind phase sc Placebo for 12 weeks. Open label extension 0.7mg/kg sc Raptiva followed by 1mg/kg/wk sc for a further 12 weeks.
  Arms: Placebo

SUMMARY:
The primary purpose of the study is to evaluate the safety and efficacy of Raptiva® compared to placebo in controlling moderate to severe chronic plaque psoriasis involving palms and/or soles scoring Palmo-plantar Pustular Psoriasis Area and Severity Index (PPPASI) ≥5 in subjects that are candidates for phototherapy or systemic therapies.

The rational of the trial is that psoriasis involving palms and/or soles is a painful condition associated with fissuring, scaling and in some instances with pustulation. Because of its localization, it is a disabling condition that limits dexterity and affects social interaction, leading to compromised quality of life; and this confers additional severity to that of plaque psoriasis on the body. The therapeutic approach for palm and sole plaque-type psoriasis usually begins with topical corticosteroid treatment. If the disease reaches a certain extent, the next step involves the addition of systemic treatments. Substances like methotrexate, retinoids and cyclosporine have shown to be efficacious, but their long-term usage is often limited by toxicity. Biologic treatments for psoriasis avoid this toxicity and offer a new therapeutic approach.

The therapeutic potential of Raptiva® to treat palm and sole psoriasis refractory to systemic treatments has been described in numerous case reports and in one placebo-controlled phase IV study. However, in all cases, the number of subjects included was low, and in most cases the trials were not prospectively designed.

Since the efficacy of Raptiva® on psoriasis of palms and soles must be determined using the validated PPPASI measure, it is necessary for scientific and ethical reasons to include a placebo arm during the first 12 weeks. Finally, as the clinical response may sometimes take longer than 12 weeks, subjects must be treated and evaluated during an additional 12-week open-label extended treatment period.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion into this trial, the subjects must fulfill all of the following criteria:

1. Subjects must have moderate to severe chronic (disease history of at least 6 months from diagnosis) plaque psoriasis involving the palms and/or soles (PPPASI =/>5) at screening, and must be candidates for phototherapy and systemic therapies.
2. Subjects must be outpatients.
3. Subjects must have stable disease at study entry (i.e. no exacerbation of psoriasis during the screening period).
4. Subjects must not have received any systemic psoriasis medication at least 14 days prior to the first administration of investigational medicinal product.
5. Subjects must not have received any topical psoriasis medication at least 14 days prior to the first administration of investigational medicinal product (emollients are allowed, as well as low potency steroids to the face and/or groin).
6. Subjects must be at least 18 years old at the time that the informed consent is obtained.
7. Female subjects of childbearing potential must use an adequate method of contraception to prevent pregnancy and must agree to continue to practice adequate contraception for the duration of their participation in the study (up to the last safety follow up visit). For male subjects, it is mandatory to practice birth control during participation in the trial, as there are no data on the effect of Raptiva® on spermatogenesis. For the purposes of this trial, women of childbearing potential are defined as "All female subjects after puberty unless they are post-menopausal for at least two years, are surgically sterile or are sexually inactive." Adequate contraception is defined as two barrier methods, or one barrier method with spermicide, or an intrauterine device or use of the oral female contraceptive.
8. Subjects must have discontinued all biological agents at least 3 months prior to the first study treatment injection.
9. Subjects must have discontinued any investigational drug or treatment at least 3 months prior to study Day 0 and/or as per washout requirements from previous protocol.
10. Subjects must be willing and able to comply with the protocol requirements for the duration of the study.
11. Subjects must have provided their written informed consent, prior to any study-related procedure not part of normal medical care, with the understanding that consent

Exclusion Criteria:

To be eligible for inclusion in this trial, the subjects must not meet any of the following criteria:

1. Hypersensitivity to Raptiva®/matching placebo or to any of their excipients.
2. Current use of any prohibited therapy (systemic or topical treatments for psoriasis, such as retinoids; immunosuppressive drugs such as methotrexate, cyclosporine A, azathioprine, or mycophenolate mofetil, or any other experimental drug).
3. Previous or current exposure to Raptiva®.
4. History of or ongoing alcohol or drug abuse.
5. History of or ongoing opportunistic infection or other serious infection. This includes any infections from the following list: Pneumocystis carinii, cytomegalovirus organ infections, Candida albicans (excluding simple localised muco-cutaneous infections), mycobacterium infections, Cryptococcus neoformans, Toxoplasma gondii, herpes simplex (excluding localised oral or genital muco-cutaneous infection), herpes zoster (excluding simple shingle eruption), cryptosporidium, Isospora belli, coccidioidomycosis, aspergillosis, histoplasmosis, and nocardiosis. This also includes diagnoses requiring more than 2 weeks of therapy, such as endocarditis and osteomyelitis treated in the past 6 months. In addition, if the subject is currently receiving antibiotics, antivirals, or antifungals for an infection or for suppression of or prophylaxis for any diagnosis, the subject will be excluded.
6. Seropositivity for hepatitis B antigen, hepatitis C antibody, or human immunodeficiency virus (HIV). Subjects will undergo testing during screening; any subjects who are found to be seropositive for hepatitis B antigen, hepatitis C antibody, or HIV will be excluded, and proper diagnosis and further therapy will be recommended.
7. Presence of active tuberculosis.
8. Presence or history of malignancy including lymphoproliferative disorders.
9. Pregnancy or breast-feeding.
10. History of hepatic cirrhosis, regardless of cause or severity.
11. History or presence of thrombocytopenia, haemolytic anaemia, clinically significant anaemia, a white blood cell count <4,000 cells/μL or >14,000 cells/μL, a haematocrit (HCT) <30%, a haemoglobin (Hgb) level <11 g/dL, or a platelet count <150,000 cells/μL.
12. Hepatic enzyme levels =/>3 times the upper limit of normal or serum creatinine level =/>2 times the upper limit of normal.
13. Vaccination with a live or live-attenuated vaccine within the 14 days prior to the first dose of investigational medicinal product.
14. Any medical condition that, in the judgment of the Investigator, would jeopardise the subject's safety following exposure to investigational medicinal product (Raptiva® or placebo equivalent) or would significantly interfere with the subject's ability to comply with the provisions of this protocol.
15. Other specific forms of psoriasis like guttate, erythrodermic or pustular psoriasis as sole or predominant form of psoriasis.
16. Immunodeficiencies.
17. Signs and symptoms suggestive of transmissible spongiform encephalopathy or family history of such.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-09; Primary Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Selenko-Gebauer, MD, Study Director — Merck Serono S.A., Geneva

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first subject's first visit: 29 Sep 2008 Date of last subject's last visit: 25 May 2009 Subjects were screened at 3 centers in Australia, of which 2 centers enrolled subjects.
  It was planned to conduct the trial in centers in Australia and Latin America; however, the trial was terminated before most centers were initiated.
Pre-assignment Details: Screening was performed within 2 weeks prior to starting trial treatment.
Period: Overall Study
Arm/Group | Raptiva | Placebo
Started | 5 | 1
Completed | 0 | 0
Not Completed | 5 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Early study termination by sponsor | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raptiva | Placebo | Total
Number analyzed (Participants) | 5 | 1 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 1 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  Australia | 5 | 1 | 6
Negative Serum Pregnancy Test [Number; unit: participants] — Participants with negative serum human chorionic gonadotrophin pregnancy test
  participants
    Negative test | 1 | 0 | 1
    Not tested (Male or surgically sterile female) | 4 | 1 | 5
Negative Urinary Pregnancy Test [Number; unit: participants] — Participants with negative urinary human chorionic gonadotrophin pregnancy test
  participants
    Negative test | 1 | 0 | 1
    Not tested (Male or surgically sterile female) | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Palmoplantar Pustular Psoriasis Area and Severity Index (PPPASI)
Description: Minimum possible score 0, maximum possible score 72.
Time Frame: Measured at Screening, Day 0, Day 7, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Population: Results not analysed due to early termination of the study
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Static Physician Global Assessment Hands and Feet (sPGA - H&F)
Description: Minimum possible score 0, maximum possible score 4.
Time Frame: Measured at Screening, Day 0, Day 7, Week 4, Week 8, Week 12, Week 16, Week 20 visits and Early Termination Visit
Population: Results not analysed due to early termination of the study
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Psoriasis Area and Severity Index (PASI)
Description: Minimum possible score 0, maximum possible score 72.
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Population: Results not analysed due to early termination of the study
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Static Physician Global Assessment (SPGA)
Description: The global response of all psoriatic lesions to therapy compared with the baseline condition using Study Day 0 Body Diagrams will be evaluated using the following categories: Cleared (100% improvement), Excellent (75-99 improvement), Good (50-74% improvement), Fair (25-49% improvement), Slight (1-24% improvement), Unchanged, or Worse
Time Frame: Measured at Screening, Day 0 and Day 7
Population: Results not analysed due to early termination of the study
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Dynamic Physician's Global Assessment of Change (dPGA)
Description: as for outcome 4
Time Frame: Measured at Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Population: Results not analysed due to early termination of the study
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Participants With Direct Physical Examination Abnormalities
Description: Physical examination included Lymph node palpation, Abdominal palpation, Auscultation of the lung, heart and intestinum
Time Frame: Measured at at screening, Day 0, Week 4, Week 12, and Early Termination visits
Population: Results not analysed due to early termination of the study
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Complaint Directed Physical Examinations
Description: Number of participants undergoing complaint directed physical examinations
Time Frame: Measure at (Day 0, Day 7, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits)
Population: Results not analysed due to early termination of the study
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Heart Rate
Time Frame: Measure at Day 0, Day 7, Week 8, Week 16 and Follow Up and Early Termination visits
Population: Results not analysed due to early termination of the study
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Arterial Blood Pressure
Time Frame: Measure at Day 0, Day 7, Week 8, Week 16 and Follow Up and Early Termination visits
Population: Results not analysed due to early termination of the study
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Temperature
Time Frame: Measure at Day 0, Day 7, Week 8, Week 16 and Follow Up and Early Termination visits
Population: Results not analysed due to early termination of the study
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Weight Measurements
Time Frame: Measured at Screening, Day 0, Day 7, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Population: Results not analysed due to early termination of the study
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Haematology Laboratory Assessments - Haemoglobin
Description: Participants with abnormal laboratory values considered by the Investigator to be clinically significant reported as adverse events.
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Subjects without values reported as adverse events | 5 | 1
  Subjects with values reported as adverse events | 0 | 0

13. Secondary Outcome: Haematology Laboratory Assessments - Haematocrit
Description: as for outcome 12
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Subjects without values reported as adverse events | 5 | 1
  Subjects with values reported as adverse events | 0 | 0

14. Secondary Outcome: Haematology Laboratory Assessments - Red Cell Count
Description: as for outcome 12
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Subjects without values reported as adverse events | 5 | 1
  Subjects with values reported as adverse events | 0 | 0

15. Secondary Outcome: Haematology Laboratory Assessments - White Cell Count
Description: as for outcome 12
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Subjects without values reported as adverse events | 5 | 1
  Subjects with values reported as adverse events | 0 | 0

16. Secondary Outcome: Haematology Laboratory Assessments - Platelets
Description: as for outcome 12
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Subjects without values reported as adverse events | 5 | 1
  Subjects with values reported as adverse events | 0 | 0

17. Secondary Outcome: Haematology Laboratory Assessments - Neutrophils
Description: as for outcome 12
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Subjects without values reported as adverse events | 5 | 1
  Subjects with values reported as adverse events | 0 | 0

18. Secondary Outcome: Haematology Laboratory Assessments - Lymphocytes
Description: as for outcome 12
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Subjects without values reported as adverse events | 5 | 1
  Subjects with values reported as adverse events | 0 | 0

19. Secondary Outcome: Haematology Laboratory Assessments - Monocytes
Description: as for outcome 12
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Subjects without values reported as adverse events | 5 | 1
  Subjects with values reported as adverse events | 0 | 0

20. Secondary Outcome: Haematology Laboratory Assessments - Eosinophils
Description: as for outcome 12
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Subjects without values reported as adverse events | 5 | 1
  Subjects with values reported as adverse events | 0 | 0

21. Secondary Outcome: Haematology Laboratory Assessments - Basophils
Description: as for outcome 12
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Subjects without values reported as adverse events | 5 | 1
  Subjects with values reported as adverse events | 0 | 0

22. Secondary Outcome: Clinical Chemistry Laboratory Assessments - Sodium
Description: as for outcome 12
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Subjects without values reported as adverse events | 5 | 1
  Subjects with values reported as adverse events | 0 | 0

23. Secondary Outcome: Clinical Chemistry Laboratory Assessments - Potassium
Description: as for outcome 12
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Subjects without values reported as adverse events | 5 | 1
  Subjects with values reported as adverse events | 0 | 0

24. Secondary Outcome: Clinical Chemistry Laboratory Assessments - Urea
Description: as for outcome 12
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Subjects without values reported as adverse events | 5 | 1
  Subjects with values reported as adverse events | 0 | 0

25. Secondary Outcome: Clinical Chemistry Laboratory Assessments - Creatinine
Description: as for outcome 12
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Subjects without values reported as adverse events | 5 | 1
  Subjects with values reported as adverse events | 0 | 0

26. Secondary Outcome: Clinical Chemistry Laboratory Assessments - Total Bilirubin
Description: as for outcome 12
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Subjects without values reported as adverse events | 5 | 1
  Subjects with values reported as adverse events | 0 | 0

27. Secondary Outcome: Clinical Chemistry Laboratory Assessments - Total Protein
Description: as for outcome 12
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Subjects without values reported as adverse events | 5 | 1
  Subjects with values reported as adverse events | 0 | 0

28. Secondary Outcome: Clinical Chemistry Laboratory Assessments - Calcium
Description: as for outcome 12
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Subjects without values reported as adverse events | 5 | 1
  Subjects with values reported as adverse events | 0 | 0

29. Secondary Outcome: Clinical Chemistry Laboratory Assessments - Aspartate Transaminase
Description: as for outcome 12
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Subjects without values reported as adverse events | 5 | 1
  Subjects with values reported as adverse events | 0 | 0

30. Secondary Outcome: Clinical Chemistry Laboratory Assessments - Alanine Transaminase
Description: as for outcome 12
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Subjects without values reported as adverse events | 5 | 1
  Subjects with values reported as adverse events | 0 | 0

31. Secondary Outcome: Clinical Chemistry Laboratory Assessments - Gamma Glutamyl Transpeptidase
Description: as for outcome 12
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Subjects without values reported as adverse events | 5 | 1
  Subjects with values reported as adverse events | 0 | 0

32. Secondary Outcome: Clinical Chemistry Laboratory Assessments - Alkaline Phosphatase
Description: as for outcome 12
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Subjects without values reported as adverse events | 5 | 1
  Subjects with values reported as adverse events | 0 | 0

33. Secondary Outcome: Clinical Chemistry Laboratory Assessments - C Reactive Protein
Description: as for outcome 12
Time Frame: Measured at Screening, Day 0, Week 4, Week 8, Week 12, Week 16, Week 20, and Early Termination visits
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Subjects without values reported as adverse events | 5 | 1
  Subjects with values reported as adverse events | 0 | 0

34. Secondary Outcome: Negative Serum Human Chorionic Gonadotrophin (hCG) Pregnancy Test
Description: A serum human chorionic gonadotrophin (hCG) pregnancy test will be conducted for all female subjects of childbearing potential prior to entering the study.
Time Frame: Measured at screening (Day -14 to Day -1)
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Negative test | 1 | 0
  Not tested (Male or surgically sterile female) | 4 | 1

35. Secondary Outcome: Negative Urinary Human Chorionic Gonadotrophin (hCG) Pregnancy Test
Description: A urinary human chorionic gonadotrophin (hCG) pregnancy test will be conducted for all female subjects of childbearing potential prior to entering the study.
Time Frame: Measured at screening (Day -14 to Day -1)
Measure: Number; unit: participants
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 5 | 1
participants
  Negative test | 1 | 0
  Not tested (Male or surgically sterile female) | 4 | 1

ADVERSE EVENTS:
Time Frame: Up to 32 weeks
Arm/Group | Raptiva | Placebo
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/1
Other Adverse Events (participants affected / at risk) | 5/5 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raptiva (N=5) | Placebo (N=1)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raptiva (N=5) | Placebo (N=1)
Flu-like symptoms (Infections and infestations) | 1 (1) | 0 (0)
Anxiety attack (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (3) | 0 (0)
Folliculitis of groin (Infections and infestations) | 1 (1) | 0 (0)
Intertrigo of groin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Left eye redness (Eye disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (6) | 0 (0)
Generalized body ache (General disorders) | 1 (1) | 0 (0)
Swelling of left heel (General disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Secondary infection, both feet (Infections and infestations) | 1 (1) | 0 (0)
Contact dermatitis, both feet (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Maculopapular rash on body (id reaction) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bilateral arm aches (nonspecific) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flu-like symptoms (General disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (3) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Infected right foot (Infections and infestations) | 1 (1) | 0 (0)
Widespread eczematous rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Telogen effluvium (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczematous rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cellulitis right leg (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other